CLINICAL TRIAL: NCT02569944
Title: Evaluation of Feasibility of Urine Collection Using Perineal Bag Versus Bladder Stimulation in Infants Less Than 12 Months Old
Brief Title: Feasibility of Bladder Stimulation in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, ROBERTO VELASCO, MD PhD, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PEDHURH-001
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- perineal bag (Active Comparator): Perineal bag was placed in infants to collect an urine sample.
  Interventions: Procedure: Perineal bag
- Bladder stimulation (Experimental): Bladder stimulation technique was used in infants of this arm to obtain an urine sample
  Interventions: Procedure: Bladder stimulation

INTERVENTIONS:
Procedure: Bladder stimulation — Patients included in this arm were stimulated to collect urine with bladder stimulation technique. This technique consists in a tapping movement in the suprapubic area, followed by a circular massage in sacral zone. This sequence lasts one minute and it is repeated five times.
  No other procedure, drug or device was done/used in this patients.
  Arms: Bladder stimulation
Procedure: Perineal bag — Patients included in this arm were placed a perineal bag to collect urine sample. No other procedure, drug or device was done/used in this patients.
  Arms: perineal bag

SUMMARY:
Randomize trial by including patients up to 12 months old in whom a urine sample by a non-sterile method was requested under physician criteria. Intention-to-treat analysis was made.

Urine dipstick was considered as altered if it was positive in leukoesterase test (≥2+) or nitrite test. In patients with an altered urine dipstick, a sterile sample was obtained for culture. If there was an initial altered urine dipstick with a subsequent negative urine culture it was considered as contaminated urine.

DETAILED DESCRIPTION:
Randomised not-blind trial developed between june 1st, 2013 and December 31st, 2014 at the Pediatric Emergency Department (PED) of Rio Hortega Universitary Hospital, a secondary hospital located in Valladolid (Spain).

Participants were infants up to one-year-old in whom a urine sample by a non-sterile method was requested under physician criteria and a written consent was signed by parents/caregivers.

The study obtained the approval of Western Valladolid Review Board.

Exclusion criteria:

Patients were excluded from the study if they met at least one of the following criteria: a) patients in whom a urine sample obtained by sterile method was needed by protocol (i.e. febrile infants less than 3 months old), b) patients with underlying disease unable to oral intake of liquids, c) patients whom parents/caregivers refused to sign the informed consent.

Randomization process:

Patients were assigned to one of the 2 groups of treatment (BS vs. PB) following a 1:1 ratio randomization sequence generated by one of the investigators (RV) using Stata® 12. (Stata Corp, College Station, Texas). After being generated, the sequence was introduced in opaque envelopes sequentially numbered.

Design of the study When, under physician criteria, it was decided to obtain a urine sample by a non-sterile method and the nurse staff that participates in the study were present at the shift, informed consent was asked to parents/caregivers. Once the consent was signed, the nurse opened the corresponding envelope, and the patient was assigned to one of the groups.

For each participant, the nurse that developed the technique filled a spreadsheet with data of the patient. Time was measured by using a stopwatch (the same one for all patients) that was not used for any purpose but the study. Urine sample was sent to the laboratory where one analyst performed the leukocyte-esterase and nitrite test. The analyst has no knowledge about the technique used on each patient and the result of the urine culture was obtained from hospital database.

If urine dipstick result was altered, another urine sample was obtained by sterile method, and urine dipstick and culture was done from that sample. Sterile sample was not routinely obtained from patients in whom non-sterile sample dipstick was normal.

In those patients who were considered as failure, the decision of obtaining an urine sample by the alternative technique, or by urethral catheterization was up to the physician who was attending the patient.

ELIGIBILITY:
Inclusion Criteria:

* infants up to one-year-old in whom a urine sample by a non-sterile method was requested under physician criteria and a written consent was signed by parents/caregivers.

Exclusion Criteria:

* patients in whom a urine sample obtained by sterile method was needed by protocol (i.e. febrile infants less than 3 months old)
* patients with underlying disease unable to oral intake of liquids
* patients whom parents/caregivers refused to sign the informed consent.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Urine sample collection | 5400 seconds
  Primary outcome is the obtention of an urine sample within the time determinate for each technique. Bladder stimulation technique is a procedure that lasts 5 minutes (300 seconds). If urine sample was obtained of patients that underwent this technique, it was considered a success. if not, a failure.
  The same was determined for the perineal bag group. In this case, our hospital's protocol recommends to use a perineal bag no longer than 30 minutes, due to risk of contamination, and after three attempts, to consider other options, so in the patients that a perineal bag was placed, if obtaining a urine sample within 90 min (5400 seconds) was considered a success. Otherwise, it was considered as a failure.
  For the purpose of the primary objective of the study, rate of falilures of each technique was compared.